CLINICAL TRIAL: NCT01386645
Title: Effect of Dietary Glycemic Index on Beta-cell Function
Acronym: GIdiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R01DK092568-01 (NIH)
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Impaired Glucose Tolerance; Oxidative Stress; Prediabetes; Impaired Fasting Glucose
Keywords: impaired glucose tolerance; prediabetes; dietary glycemic index; beta-cell function; insulin secretion; oxidative stress; glycemic variability
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State | interventions — Diet; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low GI diet (Active Comparator): low glycemic index diet
  Interventions: Other: low glycemic index (LGI) diet
- High GI diet placebo (Placebo Comparator): high glycemic index diet plus placebo
  Interventions: Other: high glycemic index (HGI) diet plus placebo (PLAC)
- High GI diet NAC (Active Comparator): high glycemic index diet plus N-acetylcysteine
  Interventions: Drug: high glycemic index diet plus N-acetylcysteine

INTERVENTIONS:
Other: low glycemic index (LGI) diet — Following a 2 week medium glycemic index control diet (glycemic index 50-55), subjects will be provided with a weight stable low glycemic index diet (glycemic index <35) for 4 weeks with all food provided by the Human Nutrition Lab
  Other Names: LGI
  Arms: Low GI diet
Other: high glycemic index (HGI) diet plus placebo (PLAC) — Following a 2 week medium glycemic index control diet (glycemic index 50-55), subjects will be provided with a weight stable high glycemic index diet (glycemic index >70) for 4 weeks, all food provided by the Human Nutrition Lab. They will take placebo capsules (matching for active N-acetylcysteine (NAC) in arm 3) twice daily for the 4 weeks on the high GI diet. The NAC vs. placebo arms (arms 2 and 3) will be double-blinded.
  Other Names: HGI/PLAC
  Arms: High GI diet placebo
Drug: high glycemic index diet plus N-acetylcysteine — Following a 2 week medium glycemic index control diet (glycemic index 50-55), subjects will be provided with a weight stable high glycemic index diet (glycemic index >70) for 4 weeks, all food provided by the Human Nutrition Lab. They will take N-acetylcysteine (NAC) two 600 mg capsules twice daily for the 4 weeks on the high GI diet. The NAC vs. placebo arms (arms 2 and 3) will be double-blinded.
  Other Names: Diet; N-acetylcysteine; NAC
  Arms: High GI diet NAC

SUMMARY:
The study will determine if increasing the highs and lows of blood glucose levels (glycemic variability) impairs insulin secretion in people with impaired glucose tolerance and/or impaired fasting glucose who are at risk for developing type 2 diabetes. Furthermore, the study will determine whether changes in beta-cell function are associated with glycemic variability and whether they are mediated by oxidative stress. To decrease or increase glycemic variability the study will provide subjects with special diets containing either low or high glycemic index foods respectively for 4 weeks. To determine if oxidative stress is a mediator, subjects on the high glycemic index diet will take either placebo or the anti-oxidant N-acetylcysteine. The study will address the hypothesis that increased glycemic variability results in increased oxidative stress and thereby exacerbates beta-cell dysfunction in individuals with impaired glucose tolerance and/or impaired fasting glucose. The findings may have important implications for the development of effective strategies aimed at the prevention and treatment of type 2 diabetes. In addition, understanding the contribution of dietary glycemic index to beta-cell dysfunction in subjects with pre-diabetes may have a significant public health impact, including changes to dietary counseling and promotion of healthier eating patterns.

DETAILED DESCRIPTION:
Type 2 diabetes is a major health problem in the United States affecting millions of people. It is caused by failure of the pancreatic beta-cells to secrete enough insulin resulting in high blood glucose levels. People with impaired glucose tolerance (IGT) and impaired fasting glucose have elevated glucose levels and are at increased risk for progressing to type 2 diabetes. The long-term objectives of this research are to better understand the factors that contribute to the loss of beta-cell function and impaired insulin secretion. High glucose levels have been shown to impair beta-cell function by causing oxidative stress, and oscillating high glucose levels increase oxidative stress even more than continuous high glucose. Diets containing foods with a high glycemic index (GI) increase the glycemic load (GL) of the diet and post-prandial glucose levels. Therefore, high GL (HGL) diets could be potentially damaging to the beta-cell by increasing glucose fluctuations and oxidative stress. Conversely, low GL (LGL) diets may be beneficial. The study explores the hypothesis that increased glycemic variability results in increased oxidative stress and thereby exacerbates beta-cell dysfunction in people with pre-diabetes.

Specific Aim 1: Determine if a HGL diet worsens and a LGL diet improves beta-cell function compared to a baseline control diet in subjects with pre-diabetes.

Specific Aim 2: Determine if increased glycemic variability on the HGL diet is associated with decreased beta-cell function and conversely if decreased glycemic variability on the LGL diet is associated with improved beta-cell function in subjects with pre-diabetes.

Specific Aim 3: Determine if oxidative stress induced by a HGL diet mediates decreases in beta-cell function by determining if 1) systemic markers of oxidative stress are associated with beta-cell function; 2) if the relationship between glycemic variability and beta-cell function is at least partially explained by oxidative stress; and 3) the anti-oxidant N-acetylcysteine (NAC) prevents decreases in beta-cell function on a HGL diet.

Study design: The study will be a randomized, parallel-design feeding study in men and women with pre-diabetes. Subjects will be randomly assigned to one of 3 separate arms (n=20/arm): 1) 4 weeks on a LGL diet (GI<35); 2) 4 weeks on a HGL diet (GI>70) + placebo twice daily; or 3) 4 weeks on a HGL diet (GI>70) + NAC 1200 mg twice daily. Subjects will be studied after a 2 week baseline control diet with a moderate glycemic load (GI 55-58) for comparison and all diets will be weight stable with the same macronutrient composition (55% carbohydrate/30% fat/15% protein). Beta-cell function will be assessed by both a frequently sampled intravenous glucose tolerance test and a meal test. Glycemic variability will be assessed by a Continuous Glucose Monitoring System and glycemic control by fructosamine. Markers of oxidative stress will be measured.

ELIGIBILITY:
Inclusion Criteria:

* impaired glucose tolerance (2 hour glucose 140-200 mg/dl after a standard 75 grams oral glucose tolerance test [OGTT]) or
* fasting glucose 100-115 mg/dl and 2 hour glucose > 100 mg/dl after a standard OGTT

Exclusion Criteria:

* diabetes or taking diabetes medications
* fasting glucose >115 mg/dl
* alanine aminotransferase (ALT) >1.5 times the upper limit of normal
* hematocrit <33%
* serum creatinine >1.5 men or >1.3 women
* multiple food allergies or intolerances
* other serious medical or inflammatory conditions
* pregnancy or lactation
* smoke or use tobacco
* take medications that affect insulin sensitivity and secretion (niacin, diabetes medications or glucocorticoids) or inflammation (anti-inflammatories such as ibuprofen, naprosyn, aspirin)
* significant gastroesophageal reflux (heartburn), swallowing problems or stomach ulcers, including those taking medication for these indications
* taking or having taken another investigational drug within the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-07; Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina M Utzschneider, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Low GI Diet: low glycemic index diet
  low glycemic index diet: Following a 2 week medium glycemic index control diet (glycemic index 50-55), subjects will be provided with a weight stable low glycemic index diet (glycemic index <35) for 4 weeks with all food provided by the Human Nutrition Lab
- High GI Diet Placebo: high glycemic index diet plus placebo
  high glycemic index diet plus placebo: Following a 2 week medium glycemic index control diet (glycemic index 50-55), subjects will be provided with a weight stable high glycemic index diet (glycemic index >70) for 4 weeks, all food provided by the Human Nutrition Lab. They will take placebo capsules (matching for active N-acetylcysteine (NAC) in arm 3) twice daily for the 4 weeks on the high GI diet. The NAC vs. placebo arms (arms 2 and 3) will be double-blinded.
Period: Overall Study
Arm/Group | Low GI Diet | High GI Diet Placebo | High GI Diet NAC
Started | 18 | 19 | 19
Completed | 18 | 18 | 17
Not Completed | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low GI Diet | High GI Diet Placebo | High GI Diet NAC | Total
Number analyzed (Participants) | 18 | 18 | 17 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (7.0) | 50.6 (10.3) | 51.2 (11.0) | 53.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 10 | 27
  Male | 10 | 9 | 7 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 8 | 14
  White | 13 | 11 | 7 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 17 | 53
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.5 (4.7) | 32.4 (6.4) | 32.7 (8.0) | 32.5 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Disposition Index
Description: The disposition index generated from an intravenous glucose tolerance test (insulin sensitivity x the acute insulin response to intravenous glucose) is a measure of beta-cell function.
Time Frame: 4 weeks
Population: 1 participant in the LGI group ate before the second IVGTT and was excluded. One participant in the HGI/PLAC group could not get a second IV and we were unable to perform the IVGTT.
Measure: Median (95% Confidence Interval); unit: unitless
Arm/Group | Low GI Diet | High GI Diet Placebo | High GI Diet NAC
Number analyzed (Participants) | 17 | 17 | 17
unitless | 708 [618 to 1244] | 793 [594 to 1257] | 791 [689 to 1215]

2. Secondary Outcome: Urine F2alpha Isoprostanes
Description: Fasting urine F2alpha isoprostane/Cr ratio. Urine isoprostanes were measured by ELISA (Oxford Biomedical Research).
Time Frame: 4 weeks
Population: Adults with prediabetes after 4 weeks on study interventions.
Measure: Median (95% Confidence Interval); unit: ng/mg
Arm/Group | Low GI Diet | High GI Diet Placebo | High GI Diet NAC
Number analyzed (Participants) | 18 | 18 | 17
ng/mg | 2.51 [1.94 to 3.81] | 3.35 [2.35 to 6.40] | 3.43 [2.53 to 6.67]

3. Secondary Outcome: Glycemic Variability
Description: Glycemic variability as measured by the standard deviation (SD) of the glucose levels from the iPro continuous glucose monitoring system (CGMS)
Time Frame: 4 weeks
Population: Adults with prediabetes with useable iPro CGMS data after the 4 week intervention.
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Low GI Diet | High GI Diet Placebo | High GI Diet NAC
Number analyzed (Participants) | 16 | 17 | 16
mg/dl | 14.20 (1.03) | 19.67 (1.57) | 17.69 (1.56)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Participants were asked about any problems related to their general health, heart, lungs, gastrointestinal system, neurologic system, urinary system and musculoskeletal system at the screening visit and at the end of the control and intervention diets using a systematic screening form. Adverse events were also reported by participants as they occurred.
Arm/Group | Low GI Diet | High GI Diet Placebo | High GI Diet NAC
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 1/18 | 1/18 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low GI Diet (N=18) | High GI Diet Placebo (N=18) | High GI Diet NAC (N=17)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Participant did not perform proper food handling and developed food poisoning with acute nausea, vomiting and diarrhea.
cracked tooth (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Participant reported that he cracked a tooth while eating broccoli that he said had something hard in it.

LIMITATIONS AND CAVEATS:
Some of the iPro CGMS devices failed to record or were dislodged. Thus, the number of participants with useable data for the CGMS variability data is less than the total enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT01386645/Prot_SAP_000.pdf